CLINICAL TRIAL: NCT04384406
Title: Assessment of the Consequences of the Abrupt Interruption of Physical and Rehabilitation Medicine Consultations During the Quarantine Period in France Between 2020 March 17th and May 11th
Brief Title: COVID-19 Outbreak Consequences for Outpatients Followed in PRM
Acronym: Handicall
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0262
Record Dates: First submitted 2020-05-10; First posted 2020-05-12 (Actual); Last update posted 2020-05-21 (Actual); Status verified 2020-05

CONDITIONS: Chronic Disabling; COVID-19
Keywords: Medical consultation; Disability; Loss of chance; Physical and Rehabilitation medicine; Home-based rehabilitation; Telehealth
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Objectives This survey aims at reporting the immediate impact of the COVID-19 epidemic on outpatients followed in Physical and Rehabilitation Medicine (PRM). It focuses on the disruption of PRM healthcare services during the quarantine period in France between 2020 March 17th and May 11th and on its medical consequences.

Method This observational study was conducted in the PRM department of a French University Hospital. Outpatients whose PRM medical consultation had been cancelled were contacted by phone between April 9th, 2020 and May 7th, 2020. A structured questionnaire was fulfilled for each patient.

Demographical and medical data were recorded, including the disabling diseases motivating the PRM outpatients' follow-up. The necessity to perform an immediate phone consultation or to schedule an urgent consultation within the next 3 weeks constituted the main judgment criterion. Other recorded criteria were: the reason for this urgent need of a medical consultation, the access to other medical services during the quarantine period, the interruption of home-based rehabilitation services and its perceived consequences for the patients.

DETAILED DESCRIPTION:
The PRM Department of Montpellier University Hospital usually provides between 8500 and 9500 medical consultations/year. A total of 830 medical consultations have been cancelled during the lockdown for COVID-19 between March 17th, 2020, and May 11th, 2020. This survey was approved by the local Institutional Review Board (IRB accreditation number: 19871).

Procedure Phone calls were performed by residents. These young doctors worked in the PRM Department for 4 months before the beginning of the outbreak and were used to the PRM medical practices of the senior practitioners. They received a special dedicated education before they start calling the patients. They fulfilled a structured questionnaire for each patient. Each resident was supervised by a senior MD. A personalized daily appointment was organized with the group of residents to check for difficulties in recording the data and to answer any question from them. Questionnaires were collected each day and data were daily implemented in a dedicated database.

Data recorded Descriptive data concerning age, description of the underlying disease, and delay from the cancelled consultation were recorded at the beginning of the call.

The main Judgment criterion is the necessity to schedule a medical consultation within the next 3 weeks: immediate telephone consultation for urgent but easy situations (like refilling a prescription or advising the patient), or short-term consultation within the next three weeks. Other patients have been proposed for a delayed consultation within the next 3 months.

Secondary objectives are: 1/ the reason for this urgent need of a medical consultation within the next 3 weeks, 2/ the category of patients for whom this need was the most prevalent, 3/the relationship between the date of the cancelled consultation and the feeling of emergency for reprogramming it, 4/ the disruption of home-based or community-based rehabilitation and its consequences for patients, and 5/ the access to other medical services for those patients during the quarantine period.

ELIGIBILITY:
Inclusion criteria:

- All outpatients whose medical appointment had been cancelled between March 17th and May 11th 2020 were contacted by phone between April 9th and May 7th 2020.

Exclusion criteria:

* Patients who had spontaneously called the hospital to ask for reprogramming the cancelled consultation before being contacted
* Patients followed by the three senior MD who preferred to call patients by themselves and who didn't want to fulfill the questionnaires for personnel reasons
* Patient who didn't answer after three phone calls

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatients from an university hospital PRM Department
Sampling Method: Non-Probability Sample
Enrollment: 467 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-05-09 (Actual)

PRIMARY OUTCOMES:
Proportion of patients necessitating the scheduling of a medical consultation | 1 day (Time of the phone call)
  Proportion of patients necessitating the scheduling of a medical consultation within the next 3 weeks

SECONDARY OUTCOMES:
the reason for this urgent need of a medical consultation | 1 day (Time of the phone call)
  the reason for this urgent need of a medical consultation
the access to other medical services during the quarantine period | 1 day (Time of the phone call)
  the access to other medical services during the quarantine period
the interruption of home-based rehabilitation services | 1 day (Time of the phone call)
  the interruption of home-based rehabilitation services and its perceived consequences for the patients

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle LAFFONT, Professor, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uh Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC